CLINICAL TRIAL: NCT02074098
Title: Endotracheal Intubation Using Macintosh Laryngoscope, Glidescope, Airwayscope During Chest Compression With Adjustment Height of a Bed
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanyang University (Other)
Responsible Party: Principal Investigator, Jaehoon Oh, Clinical fellow, Hanyang University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Intubation with a bed height
Record Dates: First submitted 2014-02-20; First posted 2014-02-28 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Tracheal Intubation; Cardiac Arrest
Keywords: intubation; Cardiopulmonary resuscitation; Manikin study
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- a 65 cm bed height (Experimental): 1) Bed height : approximately 65cm (Lowest)
  Interventions: Device: Macintosh laryngoscope; Device: Glidescope; Device: Airwayscope
- a 95cm bed height (Experimental): 2) Bed height : approximately 95cm (highest)
  Interventions: Device: Macintosh laryngoscope; Device: Glidescope; Device: Airwayscope

INTERVENTIONS:
Device: Macintosh laryngoscope — Direct Laryngoscope
Device: Glidescope — Videolaryngoscope-1
Device: Airwayscope — Videolaryngoscope-2

SUMMARY:
The purpose of this study is to determine whether a bed height make an effect to endotracheal intubation with Macintosh laryngoscope, Glidescope and Airwayscope during chest compressions in- hospital simulation cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* Experience of Intubation > 50 times
* Postgraduates year 1,2,3,4 and Emergency physicians in emergency department

Exclusion Criteria:

* Wrist or low back disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2014-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
To measure a time to expose the glottis view with a laryngoscope | 1 day
To measure a time to intubate the tube with a laryngoscope | 1 day
To estimate the success rate of Intubation | 1 day
  " Failure " means that tube is inserted in esophagus and the time is over than 120 seconds

SECONDARY OUTCOMES:
To assess the grade for the glottis view with a laryngoscopy | 1 day
  Using the Cormack-Lehane Grade system

OTHER OUTCOMES:
To assess the preference for a type of laryngoscopes | 1 day
  The participant select the type of a laryngoscope if he/she performs the endotracheal intubation under the experimental situation again.

CONTACTS AND LOCATIONS:
Locations (1):
- Hanyang University Seoul Hospital, Seoul, South Korea